CLINICAL TRIAL: NCT02170246
Title: Adjunctive Therapy With Telmisartan Instituted With ART During Acute HIV Infection to Reduce the Establishment of Central Nervous System Reservoirs of HIV and Lymph Node Fibrosis [Southeast Asia Research Collaboration With Hawaii (SEARCH) 018]
Brief Title: Analysis of Telmisartan Administered With Antiretroviral Therapy (ART) in Patients With Acute HIV Infection
Acronym: SEARCH018
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); SEARCH Research Foundation (Other); University of California, San Francisco (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); University of Hawaii (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1401013214; 1R01NS084911-01 (NIH); W81XWH-11-2-0174 (Other: Henry M. Jackson Foundation Cooperative Agreement); R01MH095613 (NIH); R01MH104141 (NIH)
Record Dates: First submitted 2014-05-22; First posted 2014-06-23 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Acute HIV Infection; HIV Infections
Keywords: Acute HIV infection; Central nervous system; Antiretroviral therapy; Telmisartan; Cerebrospinal fluid
MeSH Terms: conditions — HIV Infections | interventions — Telmisartan

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiretroviral Therapy (ART) only (No Intervention): Acute HIV-infected subjects (n=7) will be randomly assigned to a group that will receive antiretroviral therapy (the current standard of care for HIV patients) for 72 weeks.
- ART + Telmisartan (Experimental): Acute HIV-infected subjects (n=14) will be randomly assigned to a group that will receive treatment with telmisartan in addition to ART. Subjects will receive 40mg telmisartan daily for 4 weeks, followed by 80mg telmisartan daily for 44 weeks, to be taken in conjunction with ART. Subjects unable to tolerate 80mg of telmisartan will be able to de-escalate to 40mg daily. After telmisartan is stopped, subjects will continue to take ART for an additional 24 weeks (total 72 weeks).
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan
  Arms: ART + Telmisartan

SUMMARY:
This research project will study whether the drug telmisartan administered in conjunction with antiretroviral therapy (ART) will help reduce nervous system infection with HIV. The investigators are studying the effect of this treatment in people who have contracted HIV infection within the past three weeks, and thus have a form of HIV called acute HIV infection. The investigators will measure biological markers of immune activation in the blood and cerebrospinal fluid to see if telmisartan may reduce the spread of HIV reservoirs in affected patients.

DETAILED DESCRIPTION:
Note regarding the primary purpose of the study: In the Study Design section, this protocol is classified as "Other", since it is specifically designed to examine the effect of telmisartan administered in conjunction with ART on the size of HIV reservoirs in the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Have protocol-defined acute HIV-1 infection
* Be part of the SEARCH 010/RV 254 study in Bangkok, Thailand
* Ability and willingness to start ART immediately after diagnosis
* Availability for follow-up for the duration of the planned study
* Systolic blood pressure ≥ 110 mmHg
* Agree to undergo lumbar puncture at weeks 0, 48 and 72
* Ability and willingness to provide informed consent. Subjects must understand the study and sign the consent form. Persons who cannot read will have the consent form read to them by a member of the study staff and may then give informed consent by using making a thumb print.

Exclusion Criteria:

* Pregnancy (current or within the last 6 months) or breastfeeding
* Uncontrolled hypertension
* Use of thiazolidinediones or other angiotensin receptor blockers class [losartan, irbesartan, olmesartan, valsartan, candesartan (washout permitted)]
* Screening laboratory values: absolute neutrophil count < 750 cells/mm3, hemoglobin <10 gm/dL creatinine clearance <30 mL/min (estimated by the Cockcroft-Gault equation using ideal body weight)
* Known renal artery stenosis
* Known cirrhosis or severe liver disease
* Unstable coronary artery disease/angina or decompensated congestive heart failure
* Any history of intolerance to any angiotensin receptor blocker
* Need for ongoing potassium supplementation
* Any contraindication to lumbar puncture such as history of bleeding diathesis or cerebral mass lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Change in level of neopterin in the cerebrospinal fluid (CSF) of patients placed on antiretroviral therapy (ART) administered in conjunction with telmisartan, versus those placed on ART only | Change from baseline to 48 weeks following ART initiation
  Neopterin is a biological marker of immune activation. Its presence in the CSF provides information on the establishment and persistence of HIV viral reservoirs within the central nervous system of HIV-positive patients.

SECONDARY OUTCOMES:
Change in levels of mast cell progenitor-1 (MCP-1), IP-10, and HIV RNA in the cerebrospinal fluid (CSF) | Change from baseline to 48 weeks following ART initiation
  Will assess CSF levels of MCP-1, IP-10, and HIV RNA. Absolute levels of these compounds will be compared between subjects on ART + telmisartan versus those on ART only.
Change in blood plasma levels of neopterin, interleukin-6, D-dimers, soluble cluster of differentiation 14 (sCD14), and soluble cluster of differentiation 163 (sCD163) | Change from baseline to 48 weeks following ART initiation
  Will assess blood plasma levels of these biomarkers in subjects on ART + telmisartan versus those on ART only.
Change in absolute concentrations and ratios with respect to creatine of choline, myoinositol, and n-acetylaspartate (NAA) in specified brain regions | Change from baseline to 48 weeks following ART initiation
  These measurements will be made using magnetic resonance spectroscopy (MRS).
Test scores on HIV neuropsychological battery | Change from baseline to 48 weeks following ART initiation
  The assessments to be used in this study have been tested for use with native Thai speakers and will be consistent with other SEARCH study tests. SEARCH employs a HIV neurocognitive battery designed to minimize cultural bias, which has been tested in Bangkok.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Spudich, MD, MA, Principal Investigator — Yale University; Jintanat Ananworanich, MD, PhD, Study Chair — U.S. Military HIV Research Program, Bethesda, Maryland; Nittaya Phanuphak, MD, PhD, Principal Investigator — Thai Red Cross AIDS Research Centre, Bangkok, Thailand
Locations (2):
- Thailand (2):
  - Chulalongkorn University Hospital, Bangkok
  - Thai Red Cross AIDS Research Centre, Bangkok

REFERENCES:
- See also: Website: South East Asia Research Collaboration with Hawaii — http://www.searchthailand.org/